CLINICAL TRIAL: NCT05322720
Title: A Phase II Clinical Study to Evaluate the Safety and Efficacy of Recombinant hLAG-3 Fusion Protein (EOC202) Injection Combined With Albumin-bound Paclitaxel in Treatment of the Patients With HR Positive, HER2 Negative Advanced Breast Cancer With Progression After Endocrine Therapy
Brief Title: HR Positive, HER2 Negative Advanced Breast Cancer With Progression After Endocrine Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taizhou EOC Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EOC202A2102
Record Dates: First submitted 2022-03-10; First posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2021-08

CONDITIONS: Solid Tumor, Adult
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EOC202 30 mg+ albumin-bound paclitaxel (100 mg/m2); (Active Comparator): One cycle of therapy is 4 weeks (28 days), the subjects in the experimental group will receive albumin-bound paclitaxel 100 mg/m2 iv drip on Day 1 (D1), D8 and D15 of each cycle, and EOC202 30 mg subcutaneously on D2 and D16 of each cycle; the subjects in the control group will receive albumin-bound paclitaxel 100 mg/m2 iv drip on D1, D8 and D15 of each cycle. The treatment will continue until progression of disease, death, intolerable toxicity, start of other antitumor therapy, withdrawal of informed consent, loss of follow-up or termination of study for other reasons, whichever comes first.
  Interventions: Biological: EOC202; Drug: albumin-bound paclitaxel
- albumin-bound paclitaxel (100 mg/m2). (Active Comparator): One cycle of therapy is 4 weeks (28 days), the subjects in the experimental group will receive albumin-bound paclitaxel 100 mg/m2 iv drip on Day 1 (D1), D8 and D15 of each cycle, and EOC202 30 mg subcutaneously on D2 and D16 of each cycle; the subjects in the control group will receive albumin-bound paclitaxel 100 mg/m2 iv drip on D1, D8 and D15 of each cycle. The treatment will continue until progression of disease, death, intolerable toxicity, start of other antitumor therapy, withdrawal of informed consent, loss of follow-up or termination of study for other reasons, whichever comes first.
  Interventions: Drug: albumin-bound paclitaxel

INTERVENTIONS:
Biological: EOC202 — EOC202 will be SC injection
  Arms: EOC202 30 mg+ albumin-bound paclitaxel (100 mg/m2);
Drug: albumin-bound paclitaxel — albumin-bound paclitaxel will be Iv injection

SUMMARY:
Primary objective:

To evaluate the progression-free survival (PFS) for EOC202 combined with albumin-bound paclitaxel versus albumin-bound paclitaxel alone in treatment of the patients with HR positive, HER2 negative advanced breast cancer (response evaluation criteria in solid tumors, RECIST 1.1);

Secondary objectives:

1. To evaluate other efficacy variables, such as objective response rate (ORR), disease control rate (DCR), clinical benefit rate (CBR) and overall survival (OS), for EOC202 combined with albumin-bound paclitaxel versus albumin-bound paclitaxel alone in treatment of HR positive, HER2 negative advanced breast cancer;
2. To evaluate the safety of EOC202 combined with albumin-bound paclitaxel;
3. To evaluate the immunogenicity of EOC202 combined with albumin-bound paclitaxel;
4. To evaluate the change level of pharmacodynamic (PD) markers (Interferon-γ, CXCL-10).

Exploratory objectives:

To explore the correlation of baseline soluble MHC-II ligands in blood (lymphocyte activation gene-3 (Lag-3) and fibrin related antigen (FGL-1)) with safety, efficacy, PD and anti-drug antibody (ADA) in subjects in EOC202 combined with albumin-bound paclitaxel group.

DETAILED DESCRIPTION:
Overall design:

This is a randomized, open, parallel-controlled study to evaluate the efficacy and safety of EOC202 combined with albumin-bound paclitaxel versus albumin-bound paclitaxel alone in treatment of the patients with HR positive, HER2 negative advanced breast cancer.

This study plans to enroll 50 patients with HR positive, HER2 negative advanced breast cancer who have progression after endocrine therapy and are suitable for taxane therapy, and these patients will be 1:1 randomized into the following two groups for treatment:

Experimental group: EOC202 30 mg+ albumin-bound paclitaxel (100 mg/m2); Control group: albumin-bound paclitaxel (100 mg/m2). One cycle of therapy is 4 weeks (28 days), the subjects in the experimental group will receive albumin-bound paclitaxel 100 mg/m2 iv drip on Day 1 (D1), D8 and D15 of each cycle, and EOC202 30 mg subcutaneously on D2 and D16 of each cycle; the subjects in the control group will receive albumin-bound paclitaxel 100 mg/m2 iv drip on D1, D8 and D15 of each cycle. The treatment will continue until progression of disease, death, intolerable toxicity, start of other antitumor therapy, withdrawal of informed consent, loss of follow-up or termination of study for other reasons, whichever comes first.

No less than 6 cycles of therapy with albumin-bound paclitaxel will be given on the premise it is tolerable by the subject. For the combined therapy, if it is judged by investigators and approved by the sponsor that albumin-bound paclitaxel needs to be discontinued permanently for toxicity, the subject can continue to receive EOC202; on the contrary, if it is judged by investigators and approved by the sponsor that EOC202 needs to be discontinued permanently for toxicity, the subject can continue to receive albumin-bound paclitaxel.

ELIGIBILITY:
Inclusion Criteria:

1. Understanding and voluntarily signing the informed consent form;
2. Female, age ≥ 18 years and <65 years;
3. Histopathologically and molecular pathologically confirmed HR positive, HER2 negative breast cancer (based on the latest test result);

   Notes:

   Positive HR is defined as positive estrogen receptor (ER), negative or positive progesterone receptor (PR) (≥1% positive stained cells will be regarded as positive receptor); Negative HER2: negative immunohistochemical (IHC) result (0, 1+), or IHC result 2+ and negative result of in situ hybridization (ISH) amplification;
4. Progression after endocrine therapy, being suitable for late-stage rescue chemotherapy, including the following conditions (meeting any one of them):

   Primary endocrine resistance: recurrence less than two years after adjuvant endocrine therapy, or progression of disease less than 6 months after late-stage 1st-line endocrine therapy. For the patients with primary endocrine resistance, no use of other systematic therapy except endocrine therapy in relapsed/progressive period (the combined use of CDK4/6 inhibitor, Everolimus or HDAC inhibitor with endocrine therapy is allowed). There were no more than 2 lines of systemic therapy for advanced disease previously.

   Secondary (acquired) endocrine resistance: recurrence more than 2 years after adjuvant endocrine therapy and within one year after discontinuation of it, or progression of disease ≥6 months after late-stage 1st-line endocrine therapy. For the patients with secondary (acquired) endocrine resistance, at least 1 line but no more than 3 lines of endocrine therapy for advanced disease are recommended (the combined use of CDK4/6 inhibitor, Everolimus or HDAC inhibitor with endocrine therapy is allowed), and the number of lines will not be calculated for adjuvant endocrine therapy. There were no more than 3 lines of systemic therapy for advanced disease previously.
5. No use of chemotherapy for recurrent/metastatic breast cancer;
6. At least one extracranial measurable lesion (RECIST 1.1);
7. Peripheral blood absolute monocyte count (AMC) <0.25×109/L (tested by local laboratory, it is allowed to be repeated once if the AMC is ranged from 0.25~0.35×109/L at screening);
8. Eastern Cooperative Oncology Group (ECOG) Performance Status score 0-1;
9. Expected survival ≥3 months;
10. Recovery of toxicity induced by previous therapy (except alopecia) to grade 1 (National Cancer Institute - Common Terminology Criteria for Adverse Events version 5.0 [NCI CTCAE v5.0]) or normal level;
11. Good organ function within 1 week prior to the first dose of study drug:

    Hematology: no transfusion of platelet or any growth factor within 7 days prior to the screening visit, white blood cell count ≥3×109/L, absolute neutrophil count (ANC) ≥1.5×109/L, platelet count ≥100×109/L, hemoglobin ≥90 g/L; Hepatic function: serum total bilirubin ≤1.5× upper limit of normal (ULN), or total bilirubin ≤3×ULN in case of Gilbert's syndrome; aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5×ULN, or AST and ALT≤5×ULN in case of hepatic metastasis; Renal function: serum creatinine ≤1.5×ULN.
12. The female subjects of childbearing potential must have negative pregnancy test within 1 week prior to the first dose of study drug, and they and their spouses agree to take effective contraceptive measures during the study and within 6 months after the last dose

Exclusion Criteria:

1. Known uncontrollable or symptomatic central nervous system metastasis, including brain metastasis or meningeal metastasis, or symptoms suggestive of cancerous meningitis, leptomeningeal disease and/or progressive growth. Patients with a history of central nervous system metastasis or spinal cord compression are allowed to be enrolled if they have received definite local treatment (e.g., radiotherapy, surgical therapy), have discontinued anticonvulsant drugs and steroids for at least 4 weeks prior to the first dose of study drug and have stable clinical manifestations;
2. Previous use of high-dose chemotherapy plus hemopoietic stem cell transplantation;
3. Grade 4 operation performed within 4 weeks prior to the first dose of study drug, or grade 2 or 3 operation performed within 7 days prior to the first dose of study drug;
4. Abnormal thyroid function that is poorly controlled after treatment;
5. Chemotherapy, endocrine therapy or treatment with other investigational product within 4 weeks or 5 half-lives prior to the first dose of study drug (whichever is longer); or radiotherapy within 2 weeks prior to the first dose of study drug (except the palliative radiotherapy for non-target lesion, enrollment will be allowed if the toxicity is resolved);
6. Serious or uncontrolled heart disease (New York Heart Association [NYHA] grade III-IV) within 6 months prior to the first dose of study drug, including myocardial infarction, severe/unstable angina pectoris, ≥grade 2 persistent arrhythmia in accordance with NCI CTCAE v5.0, atrial fibrillation of any grade, coronary/peripheral artery bypass grafting, symptomatic congestive heart failure; or presence of cerebrovascular accident, including transient ischemic attack, symptomatic pulmonary embolism, etc.;
7. Presence of other malignant tumors within 5 years prior to the first dose of study drug (except for basal cell or squamous cell carcinoma of skin, superficial bladder cancer and carcinoma in situ of cervix, which have been cured);
8. Other concomitant disease seriously hazardous to patient's safety or affecting completion of the study as judged by investigators, except for tumor;
9. Presence of one of the following conditions: active infection considered by investigators that may affect patient's participation in the study or the study results; positive hepatitis B surface antigen, and hepatitis B virus (HBV) DNA copy > ULN (patients with HBV DNA copy reduced to normal range after antiviral therapy are allowed to be enrolled); positive hepatitis C virus antibody and hepatitis C virus (HCV) RNA copy >ULN; positive human immunodeficiency virus (HIV); or any serious infection requiring systematic treatment within 4 weeks prior to the first dose of study drug;
10. Clinically significant abnormality indicated on electrocardiography (ECG), including but not limited to serious arrhythmia, prolonged QT interval (QTcF>470 ms, QTcF=QT/RR0.33); or presence of various conditions that may increase the risk of prolonged QT interval, e.g., known history of prolonged QTc, congenital long QT syndrome, Brugada syndrome, torsade de pointes, uncontrollable electrolyte disorder (e.g., calcemia, hypokalaemia and hypomagnesaemia, etc.);
11. Previous diagnosis of autoimmune disease or requiring long-term use of systemic corticosteroids (dose >10 mg/day prednisone or equivalent) or other immunosuppressants within 4 weeks prior to the first dose of study drug; however, patients are allowed to be enrolled in the following conditions: in the absence of active autoimmune disease, inhaled or topical steroids, or adrenaline replacement therapy at the dose ≤10 mg/day Prednisone equivalent is allowed to be used;
12. Treatment with systematic immunostimulatory drugs (including but not limited to interferon-α (IFN-α) and interleukin 2 (IL-2)) within 6 weeks or 5 half-lives prior to the first dose of study drug (whichever comes later);
13. Vaccination with live attenuated vaccine, protein vaccine, mRNA or DNA vaccine within 4 weeks prior to the first dose of study drug, or expected to receive the above vaccines during the study;
14. Previous allergy to macromolecular protein preparation or protein, or Quincke's edema (also known as angioneurotic edema), or known allergy to any component of the study drug;
15. History of clear mental disorder, or history of psychotropic drug abuse, drug addiction or alcohol abuse;
16. Received organ transplant;
17. Women who are pregnant or breastfeeding;
18. Having participated in any other drug clinical trial within 4 weeks prior to the first dose of study drug or currently receiving treatment in other clinical trials (except those who are participating in the follow-up of overall survival in one study);
19. Patients with other conditions that are not suitable to participate in the clinical trial, as considered by the investigator.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
PFS | up to 30 months
  To evaluate the progression-free survival (PFS)

SECONDARY OUTCOMES:
ORR | 30 months
  objective response rate (ORR)
DCR | 30 months
  disease control rate
CBR | 30 months
  clinical benefit rate
OS | 30 months
  overall survival
the safety of EOC202 combined with albumin-bound paclitaxel | 30 months
  To evaluate the safety of EOC202 combined with albumin-bound paclitaxel
The immunogenicity of EOC202 combined with albumin-bound paclitaxel; | 30 months
  o evaluate the immunogenicity of EOC202 combined with albumin-bound paclitaxel;
the change level of PD markers (Interferon-γ, CXCL-10) | 30 months
  To evaluate the change level of pharmacodynamic (PD) markers (Interferon-γ, CXCL-10)

OTHER OUTCOMES:
The correlation of baseline soluble MHC-II ligands in blood (Lag-3 and FGL-1）with safety, efficacy, PD and ADA | up to 30 months
  To explore the correlation of baseline soluble MHC-II ligands in blood (lymphocyte activation gene-3 (Lag-3) and fibrin related antigen (FGL-1)) with safety, efficacy, PD and anti-drug antibody (ADA) in subjects in EOC202 combined with albumin-bound paclitaxel group

CONTACTS AND LOCATIONS:
Overall Officials: Xichun Hu, Ph.D, Principal Investigator — Fudan University

IPD SHARING:
Plan to Share IPD: No